CLINICAL TRIAL: NCT01712360
Title: An Open-Label, Multi-Center, Multiple-Application Pharmacokinetic Study of NAFT-500 in Pediatric Subjects With Tinea Cruris and Tinea Pedis and NAFT-600 in Pediatric Subjects With Tinea Pedis
Brief Title: Pharmacokinetic Study of Pediatric Subjects With Tinea Cruris and Tinea Pedis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUS 90200/1023/0; Tinea Pedis and Cruris
Record Dates: First submitted 2012-10-16; First posted 2012-10-23 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Tinea Pedis; Tinea Cruris
Keywords: Tinea Pedis; Tinea Cruris; Athlete foot; Jock itch
MeSH Terms: conditions — Tinea Pedis; Tinea Cruris | interventions — naftifine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NAFT500 (pediatric) (Experimental): Topical once a day for two weeks
  Interventions: Drug: NAFT500 (pediatric)
- NAFT600 (pediatric) (Experimental): Topical once a day for two weeks
  Interventions: Drug: NAFT600 (pediatric)
- NAFT500 (adult) (Experimental): Topical once a day for two weeks
  Interventions: Drug: NAFT500 (adult)
- NAFT600 (adult) (Experimental): Topical once a day for two weeks
  Interventions: Drug: NAFT600 (adult)

INTERVENTIONS:
Drug: NAFT500 (pediatric) — Applied to both feet and groin area
  Other Names: NAFT500; naftifine; naftifine hydrochloride
  Arms: NAFT500 (pediatric)
Drug: NAFT600 (pediatric) — Applied to both feet only
  Other Names: NAFT600; naftifine; naftifine hydrochloride
  Arms: NAFT600 (pediatric)
Drug: NAFT500 (adult) — Applied to both feet and groin area
  Other Names: NAFT500; naftifine; naftifine hydrochloride
  Arms: NAFT500 (adult)
Drug: NAFT600 (adult) — Applied to both feet
  Other Names: NAFT600; naftifine; naftifine hydrochloride
  Arms: NAFT600 (adult)

SUMMARY:
This study is being done to see how the body is affected when a study drug is applied to both feet if the subject has athlete's foot or to both feet and the groin area if the subject has both athlete's foot and jock itch. Safety of the drug and how well the drug works will also be measured.

DETAILED DESCRIPTION:
Study population, diagnosis, and main criteria for inclusion:

Tinea pedis and Tinea cruris (NAFT-500):

Male or non-pregnant female subjects aged 12 to 17 years, 11 months old of any race with Tinea pedis and Tinea cruris infections confirmed by a positive potassium hydroxide (KOH) analysis from both the feet and bikini area. Both cases (feet and bikini area) must be characterized by clinical evidence of a Tinea pedis and Tinea cruris infection. Additional, approximately 4 pharmacokinetic (PK) evaluable adult subjects with the same condition will serve as a control.

Tinea pedis (NAFT-600):

Male or non-pregnant female subjects aged 12 to 17 years, 11 months old of any race with Tinea pedis infection confirmed by a positive potassium hydroxide (KOH) analysis from both feet. Both feet must be characterized by clinical evidence of a Tinea pedis infection. Additional, approximately 4 pharmacokinetic (PK) evaluable adult subjects with the same condition will serve as a control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have Tinea pedis on both feet and Tinea cruris infections for NAFT-500; both conditions must be characterized by clinical evidence of a Tinea infection.
* Subjects must have Tinea pedis on both feet for NAFT-600; the condition must be characterized by clinical evidence of a Tinea infection.

Exclusion Criteria:

* A known hypersensitivity to study medications or their components
* Any severe condition of Tinea pedis (incapacitating)
* Any dermatological disease and or condition in the treatment or surrounding area that may prevent application of the study product such as foot psoriasis, corns and /or callus involving any web spaces, or atopic or contact dermatitis
* Positive pregnancy test
* Any history or current evidence (physical or laboratory) of anemia

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Study Director — Merz Pharmaceutical, LLC
Locations (4):
- United States (2):
  - Merz Investigative Site #001272, Austin, Texas
  - Merz Investigative Site #001261, College Station, Texas
- Merz Investigative Site #180001, Santo Domingo, Santo Domingo Province, Dominican Republic
- Merz Investigative Site #504001, San Pedro Sula, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NAFT500 (Pediatric) | NAFT600 (Pediatric) | NAFT500 (Adult) | NAFT600 (Adult)
Started | 22 | 22 | 6 | 6
Completed | 22 | 21 | 6 | 4
Not Completed | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set which is the subset of subjects who have been exposed to the study medication at least once
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFT500 (Pediatric) | NAFT600 (Pediatric) | NAFT500 (Adult) | NAFT600 (Adult) | Total
Number analyzed (Participants) | 22 | 22 | 6 | 6 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 0 | 0 | 44
  Between 18 and 65 years | 0 | 0 | 6 | 6 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.5) | 14.7 (1.7) | 38.7 (6.5) | 31.7 (11.2) | 19.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 0 | 2 | 11
  Male | 17 | 18 | 6 | 4 | 45
Region of Enrollment [Number; unit: participants]
  United States | 0 | 7 | 6 | 6 | 19
  Honduras | 20 | 0 | 0 | 0 | 20
  Dominican Republic | 2 | 15 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Naftifine Hydrochloride Pharmacokinetics Variables, Single and Multiple Dose
Description: Variables will be derived from naftifine plasma concentration at day 1. Variables to be analyzed:
  - Partial area under the plasma concentration-time curve (0-24 hours postdose) (AUC), as calculated using the linear trapezoid rule.
  Variables will be derived from naftifine plasma concentration at day 14. Variables to be analyzed:
  - Area under the plasma concentration-time curve (AUC) within one dosing interval at steady state (SS). AUCτ,ss= Area under the concentration curve within a dosing interval (τ = 24 hours) at steady state
Time Frame: Day 1 and Day 14
Population: Pharmacokinetic analysis set (PKS), defined as the subset of subjects in the safety evaluation set (SES) with evaluable pharmacokinetic (PK) samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | NAFT500 (Pediatric) | NAFT600 (Pediatric) | NAFT500 (Adult) | NAFT600 (Adult)
Number analyzed (Participants) | 20 | 22 | 6 | 5
h*pg/mL
  AUC0-24 Day 1, Single Dose | 138262.2 (50.2) | 15890.1 (211.6) | 68634.2 (95.4) | 17213.9 (88.1)
  AUCτ,ss Day 14 Multiple Dose | 192485.4 (74.9) | 60038.5 (131.1) | 124596.0 (49.9) | 72849.8 (71.1)

2. Secondary Outcome: Efficacy Variables
Description: Efficacy variables to be analyzed after 2 weeks of once daily application of both products (NAFT-500 or NAFT-600).
  Efficacy variables to be analyzed:
  * Complete cure
  * Treatment effectiveness
  * Mycological cure
  * Clinical success
  * Clinical cure
Time Frame: Day 28
Population: Full analysis set, defined as subset of subjects in the safety evaluation set (SES) for whom any efficacy variable is available.
Measure: Number (90% Confidence Interval); unit: Percentage (%) of subjects (90% CI)
Groups:
- NAFT500 (Pediatric, Foot); NAFT500 (Pediatric, Groin): Topical once a day for two weeks
  NAFT500 (pediatric): Applied to both feet and groin area
- NAFT500 (Adult, Foot); NAFT500 (Adult, Groin): Topical once a day for two weeks
  NAFT500 (adult): Applied to both feet and groin area
Arm/Group | NAFT500 (Pediatric, Foot) | NAFT500 (Adult, Foot) | NAFT500 (Pediatric, Groin) | NAFT500 (Adult, Groin) | NAFT600 (Pediatric) | NAFT600 (Adult)
Number analyzed (Participants) | 22 | 6 | 22 | 6 | 22 | 5
Percentage (%) of subjects (90% CI)
  Complete Cure | 59.1 [39.5 to 76.7] | 0 [0 to 0] | 63.6 [43.9 to 80.4] | 16.7 [0.9 to 58.2] | 27.3 [12.6 to 46.8] | 0 [0 to 0]
  Treatment Effectiveness | 63.6 [43.9 to 80.4] | 0 [0 to 0] | 63.6 [43.9 to 80.4] | 50.0 [15.3 to 84.7] | 54.5 [35.3 to 72.9] | 20.0 [1.0 to 65.7]
  Mycological Cure | 68.2 [48.5 to 84.0] | 16.7 [0.9 to 58.2] | 72.7 [53.2 to 87.4] | 66.7 [27.1 to 93.7] | 63.6 [43.9 to 80.4] | 20.0 [1.0 to 65.7]
  Clinical Success | 90.9 [74.1 to 98.4] | 66.7 [27.1 to 93.7] | 90.9 [74.1 to 98.4] | 66.7 [27.1 to 93.7] | 81.8 [63.1 to 93.5] | 80 [34.3 to 99.0]
  Clinical Cure | 81.8 [63.1 to 93.5] | 16.7 [0.9 to 58.2] | 81.8 [63.1 to 93.5] | 33.3 [6.3 to 72.9] | 40.9 [23.3 to 60.5] | 20.0 [1.0 to 65.7]

3. Primary Outcome: Naftifine Hydrochloride Pharmacokinetics Variables, Single and Multiple Dose
Description: Variables will be derived from naftifine plasma concentration at day 1. Variables to be analyzed:
  - Maximum observed plasma concentration (Cmax): the highest plasma concentration in each subject after single dose.
  Variables will be derived from naftifine plasma concentration at day 14. Variables to be analyzed:
  - Maximum observed plasma concentration (Cmax): the highest plasma concentration in each subject at steady state (SS).
Time Frame: Day 1 and Day 14
Population: Pharmacokinetic analysis set (PKS), defined as the subset of subjects in safety evaluation set (SES) with evaluable pharmacokinetic (PK) samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | NAFT500 (Pediatric) | NAFT600 (Pediatric) | NAFT500 (Adult) | NAFT600 (Adult)
Number analyzed (Participants) | 20 | 22 | 6 | 5
pg/mL
  Cmax Day 1, Single Dose | 9213.35 (48.4) | 1397.77 (153.8) | 3983.34 (83.0) | 1741.02 (69.2)
  Cmax, SS Day 14 Multiple Dose | 12727.36 (67.2) | 3813.38 (153.9) | 6826.70 (51.3) | 3538.84 (73.3)

4. Secondary Outcome: Efficacy Variables
Description: Efficacy variables to be analyzed after 2 weeks of once daily application of both products (NAFT-500 or NAFT-600).
  Efficacy variables to be analyzed:
  - Subject satisfaction
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | NAFT500 (Pediatric, Foot) | NAFT500 (Adult, Foot) | NAFT500 (Pediatric, Groin) | NAFT500 (Adult, Groin) | NAFT600 (Pediatric) | NAFT600 (Adult)
Number analyzed (Participants) | 22 | 6 | 22 | 6 | 22 | 5
Percentage (%) of subjects
  Excellent Improvement | 81.8 | 0 | 86.4 | 16.7 | 54.5 | 20.0
  Much Improved | 13.6 | 83.3 | 13.6 | 50.0 | 36.4 | 60.0
  Improved | 4.5 | 16.7 | 0 | 33.3 | 4.5 | 20.0
  No Change | 0 | 0 | 0 | 0 | 0 | 0
  Worse | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | NAFT500 (Pediatric) | NAFT600 (Pediatric) | NAFT500 (Adult) | NAFT600 (Adult)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/22 | 2/22 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAFT500 (Pediatric) (N=22) | NAFT600 (Pediatric) (N=22) | NAFT500 (Adult) (N=6) | NAFT600 (Adult) (N=6)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No